CLINICAL TRIAL: NCT01558830
Title: Safety of Amiodarone and Ranolazine Together in Patients With Stable Angina
Brief Title: Safety of Amiodarone and Ranolazine Together in Patients With Angina
Acronym: SARA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cardiovascular Consultants of Nevada (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IN-US-259-0121
Record Dates: First submitted 2012-03-18; First posted 2012-03-20 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Chronic Stable Angina; Coronary Artery Disease; Atrial Fibrillation; Ventricular Tachycardia
Keywords: amiodarone; ranolazine; safety; arrhythmia
MeSH Terms: conditions — Angina, Stable; Coronary Artery Disease; Atrial Fibrillation; Tachycardia, Ventricular; Arrhythmias, Cardiac | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sugar pill (Placebo Comparator): one pill twice daily, uptitrated to two pills twice daily to mirror ranolazine prescription strategy
  Interventions: Drug: placebo
- Ranolazine (Active Comparator): 500 mg twice daily, titrated to 1000 mg twice daily if needed for relief of anginal symptoms
  Interventions: Drug: ranolazine

INTERVENTIONS:
Drug: ranolazine — ranolazine 500mg twice daily, may increase to 1000 mg twice daily for therapy optimization in treating chronic stable angina
  Other Names: Ranexa
  Arms: Ranolazine
Drug: placebo — one pill twice daily, to increase to two pills twice daily to mirror standard ranolazine treatment strategy
  Arms: sugar pill

SUMMARY:
Ranolazine is an effective and remarkably safe agent for the treatment of patients with chronic stable angina, but its inhibition of voltage gated potassium channels and electrocardiogram (EKG) corrected QT (QTc) prolongation properties have lead many to question its safety when combined with antiarrhythmic drugs. The investigators have proposed a study to determine the safety of ranolazine in patients with chronic stable angina who also take amiodarone. And are conducting a prospective single-center randomized single-blinded placebo controlled trial to run out of our large cardiology practice setting at Cardiovascular Consultants of Nevada. The hypothesis is that there will be no difference in the ventricular arrhythmia burden. The primary outcome will be the measurement of ventricular arrhythmia episodes on serial holter monitor and other serially acquired recordings (such as electrocardiogram, pacemaker or implantable defibrillator (ICD) data, and stress test data) over a three month trial period.

ELIGIBILITY:
Inclusion Criteria:

* ischemic cardiac disease
* chronic anginal symptoms
* on amiodarone therapy for other cardiac conditions

Exclusion Criteria:

* pregnant
* non-English speaking
* unstable angina
* baseline electrocardiogram (EKG) corrected QT (QTc)>490ms
* severe thyroid dysfunction
* heart block without a pacer system
* liver disease

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-04 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
ventricular arrhythmia | 3 months
  primary outcome is the burden of ventricular arrhythmias measured on serial holter monitor recordings, stress test recordings, pacemaker or implantable defibrillator (ICD) recordings if available, at baseline and serially to trial completion.

SECONDARY OUTCOMES:
atrial arrhythmia burden | 3 months
  burden of atrial arrhythmias will be measured on serial holter monitor recordings
Electrocardiogram (EKG) corrected QT (QTc) interval measurement | over the 3 month trial
  The electrocardiogram (EKG) corrected QT (QTc) interval be quantitated at baseline and serially to trial completion
hospitalization | 3 months
  Hospitalization rates, if any, will be serially quantitated to trial completion
syncope hospitalization | 3 months
  syncope hospitalization rate quantitation to trial completion
liver function assay | 3 months
  serum liver function testing will be conducted at baseline and serially to trial completion

CONTACTS AND LOCATIONS:
Overall Officials: Erik J SIrulnick, MD, Principal Investigator — Cardiovascular Consultants of Nevada
Locations (2):
- United States (2):
  - Cardiovascular Consultants of Nevada, Henderson, Nevada
  - Cardiovascular Consultants of Nevada, Las Vegas, Nevada